CLINICAL TRIAL: NCT01204112
Title: A Phase 1, Open Label, Fixed-Sequence Study To Estimate The Effect Of Repeat-Dose Rifampin On The Pharmacokinetics Of CP-690,550 In Healthy Volunteers
Brief Title: Estimate The Effect Of Repeat-Dose Rifampin On The Pharmacokinetics Of CP-690,550 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A3921056
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Healthy
Keywords: Drug-Drug Interaction; Tasocitinib (CP-690; 550); Rifampin; Healthy Volunteers
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tasocitinib (CP-690,550) plus Rifampin (Experimental)
  Interventions: Drug: Tasocitinib (CP-690,550) plus Rifampin

INTERVENTIONS:
Drug: Tasocitinib (CP-690,550) plus Rifampin — Period 1, Day 1: Tasocitinib (CP-690,550) 30 mg (single oral dose) as six 5 mg tablets Period 2, Day 1-7: Rifampin 600 mg (single oral dose) q24h Period 2, Day 8: Tasocitinib (CP-690,550) 30 mg (single oral dose) as six 5 mg tablets Period 2, Day 9: No treatment (discharge)

SUMMARY:
The current study is designed to estimate the effect of rifampin (600 mg orally every 24 hours for 7 days) on pharmacokinetics of single 30 mg dose (CP-690,550) in normal healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects (of non-childbearing potential)

Exclusion Criteria:

* Clinically significant disease or condition
* Recent serious infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
AUCinf of tasocitinib (CP-690,550) | 9 days
Cmax of tasocitinib (CP-690,550) | 9 days

SECONDARY OUTCOMES:
AUClast, Tmax, t1/2 of tasocitinib (CP-690,550) | 9 days
Safety: clinical laboratory abnormalities, AE reporting, and vital signs (blood pressure/pulse rate). | 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921056&StudyName=Estimate%20The%20Effect%20Of%20Repeat-Dose%20Rifampin%20On%20The%20Pharmacokinetics%20Of%20CP-690%2C550%20In%20Healthy%20Volunteers